CLINICAL TRIAL: NCT00518921
Title: Phase IIa Efficacy and Safety Trial of Capadenoson in Patients With Chronic Stable Angina
Brief Title: Capadenoson in Angina Pectoris
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12484; EudraCT 2007-000425-22
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Stable Angina
Keywords: adenosin agonist; chronic stable angina
MeSH Terms: conditions — Angina, Stable | interventions — capadenoson

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Capadenoson (BAY 68-4986)
- Arm 2 (Experimental)
  Interventions: Drug: Capadenoson (BAY 68-4986)
- Arm 3 (Experimental)
  Interventions: Drug: Capadenoson (BAY 68-4986)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capadenoson (BAY 68-4986) — 1mg Capadenoson, double dummy
  Arms: Arm 1
Drug: Capadenoson (BAY 68-4986) — 2mg Capadenoson, double dummy
  Arms: Arm 2
Drug: Capadenoson (BAY 68-4986) — 4mg Capadenoson, double dummy
  Arms: Arm 3
Drug: Placebo — Placebo, double dummy
  Arms: Arm 4

SUMMARY:
This is a multi-center and multi-national,randomized, double blind, placebo-controlled, 28-day treatment study with BAY 68-4986 taken orally or a matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* The primary diagnosis is chronic stable angina of mild-moderate intensity as defined by the Canadian Cardiovascular Society Functional Class II-III, in the presence of definitive coronary artery disease.
* Male or female subjects aged 35 to 75 years (if female, only if postmenopausal or permanently sterilized)
* Stable angina of mild-moderate intensity (Canadian class II-III) with anti-anginal medication not changed for the last 5 weeks

Exclusion Criteria:

* Inability to withdraw current anti-anginal therapy
* Inability to withdraw any concomitant therapy that would interfere with interpretation of study results

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Total exercise time | 28 days for ETT and 42 days for safety

SECONDARY OUTCOMES:
Time to angina onset | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Czechia (7):
  - Brno
  - Hodonín
  - Kroměříž
  - Olomouc
  - Ostrava
  - Pilsen
  - Prague
- Hungary (5):
  - Balatonfüred
  - Kecskemét
  - Miskolc
  - Pécs
  - Zalaegerszeg
- Israel (3):
  - Hadera, Israel
  - Rehovot, Israel
  - Safed, Israel
- Italy (4):
  - Mestre, Venezia
  - Genova
  - Pavia
  - Trieste
- Poland (11):
  - Bialystok
  - Gdansk
  - Gdynia
  - Katowice
  - Krakow
  - Legnica
  - Lodz
  - Starogard Gdański
  - Szczecin
  - Warsaw
  - Wroclaw
- Slovakia (3):
  - Bratislava
  - Nitra
  - Nové Zámky